CLINICAL TRIAL: NCT01777919
Title: A PHASE II CLINICAL TRIAL FOR THE EVALUATION OF THE EFFICACY OF DISULFIRAM/COPPER COMBINATION AS AN ADJUVANT AND CONCURRENT CHEMOTHERAPY IN THE TREATMENT OF NEWLY DIAGNOSED GLIOBLASTOMA MULTIFORM
Brief Title: Disulfiram/Copper Combination In The Treatment of Newly Diagnosed Glioblastoma Multiform
Acronym: GLIODIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Olympion Medical Center (Other)
Collaborators: University of Ioannina (Other); University of Eastern Finland (Other); University of Ulm (Other)
Responsible Party: Principal Investigator, Petros Karamanakos, MD, PhD, Neurosurgeon, MD, PhD, Olympion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK-18081973; NCT01982370 (obsolete NCT alias)
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Disulfiram; Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temozolomide+Disulfiram/copper (Experimental): Disulfiram/copper combination will be started on the 5th postoperative day and before the initiation of the standard radiochemotherapy (fractionated irradiation with a total dose of 60 Gy with concomitant 75 mg/m2 body surface temozolomide each day, including weekends, during irradiation). After completion of the radiation therapy patients will receive maintenance temozolomide 150-200 mg/m2 body surface on Days 1-5 every 28 days for 6 months. Daily administration of disulfiram and copper will take place for the whole study period.
  NOTE: Patients may receive additional maintenance temozolomide at the discretion of the treating medical oncologist.
  Interventions: Drug: Temozolomide; Drug: Disulfiram; Drug: Copper

INTERVENTIONS:
Drug: Temozolomide — already included
  Other Names: Temodar
Drug: Disulfiram — already included
  Other Names: Antabuse
Drug: Copper — already included

SUMMARY:
Glioblastoma multiform (GBM) is the most common malignant primary brain tumor in adults. Despite maximal treatment tumor relapse occurs regularly accompanied by unfavourable prognosis. Among other reasons, it is believed that this could be in part due to the existence of the so-called tumor stem cells (TSCs), a cellular subfraction within GBM which escape therapy by being highly resistant to irradiation and chemotherapy and thus constituting the source of tumor recurrence.

GBM, like many other cancers, show a sub-population of aldehyde dehydrogenase (ALDH) overexpressing TSCs. More specifically, ALDH1A1, a cytoplasmatic isoform of ALDH, proved to be a novel stem cell marker in human GBM. In addition, ALDH1A1 has been shown to be a mediator for resistance of GBM to temozolomide (TMZ) and a reliable predictor of clinical outcome; prognosis of patients with a high level of ALDH1A1 expression was poor compared with that of patients with low levels. Consequently, ALDH1A1 may serve as a potential target to improve treatment of human GBM through inhibition of the enzyme.

Disulfiram (DSF) has been used for more than sixty years in the treatment of chronic alcoholism because of the unpleasant symptoms it provokes after ethanol intake. The underlying mechanism is believed to be the accumulation of acetaldehyde in the blood, due to inhibition of the liver ALDHs. Actually, DSF is a strong inhibitor of ALDH1A1 and relatively non-toxic at therapeutic (for chronic alcoholism) doses that can penetrate the blood-brain barrier. In addition, DSF has been shown to be cytotoxic on GBM stem-like cells, inhibiting the growth of TMZ resistant GBM cells and blocking self-renewal by ~100% , while it has been identified as an inhibitor of human GBM stem cells in high-throughput chemical screens. Interestingly, a number of these actions were copper-dependent.

In the current Phase II clinical trial, DSF/copper combination will be tested as an adjunctive and concurrent chemotherapy in the treatment of newly diagnosed GBM. According to our hypothesis, initiation of DSF chemotherapy after the resection of the tumor and before the introduction of the standard radio-chemotherapy will inhibit ALDH1A1 of GBM TSCs making them more susceptible to radio-chemotherapy and possibly reducing the recurrence rate of GBM. On the other hand, the addition of copper will probably enhance the cytotoxic effects of DSF possibly through augmentation of its pro-apoptotic and proteasomal inhibitory actions.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed diagnosis of glioblastoma (World Health Organization [WHO] grade IV astrocytoma). Patients must be newly diagnosed with unifocal supratentorial GBM amenable to gross total resection (< 1 cm. enhancing rim) and not yet received chemoradiation.
2. Patient must have undergone a gross total surgical resection of the tumor mass with post-surgical MRI (performed within 72 hours after operation) demonstration of adequacy defined as < 1.0 cm of residual enhancement away from resection cavity perimeter.
3. Ability to start disulfiram on the 5th postoperative day
4. ≥ 18 years of age
5. Karnofsky Performance Status (KPS) ≥ 70%
6. Adequate bone marrow function, defined as:

   Absolute neutrophil count ≥ 1000 cells/mm3 Hemoglobin ≥ 10 g/dL Platelet count ≥ 100,000 cells/mm3
7. Adequate hepatic function, defined as:

   Bilirubin ≤ 2.0 mg/dL Alkaline phosphatase (ALP), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 4x upper limit of normal (ULN)
8. Adequate renal function, defined blood urea nitrogen (BUN) < 30 mg/dL and creatinine < 2 mg/dL
9. Prothrombin time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6x control unless therapeutically warranted
10. Female patients of child-bearing potential must have negative serum or urine pregnancy test
11. If not surgically sterile, male and female patients of childbearing age must use double barrier contraception (hormonal; intrauterine device; barrier)
12. Patient must give written informed consent prior to any study-specific procedures being implemented.

Exclusion Criteria:

1. Recurrent disease
2. Infratentorial or multifocal tumor.
3. Placement of Gliadel wafer
4. No severe, active comorbidity, including any of the following:

   * Unstable angina and/or congestive heart failure requiring hospitalization
   * Transmural myocardial infarction within the last 6 months
   * Chronic obstructive pulmonary disease
   * Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   * Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness
   * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
   * Known history of an autoimmune disorder
   * Presence of any other active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin)
5. Alcoholism
6. Breastfeeding
7. Prior or planned chemotherapy, immunotherapy, biologic therapy, radiation therapy, radioimmunotherapy, hormonal therapy, or experimental therapy for brain tumor
8. History of severe allergic reaction to contrast media.
9. Inability to undergo an MRI.
10. Patients treated on any other therapeutic clinical trial within 30 days prior to study entry or during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months

SECONDARY OUTCOMES:
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Petros N Karamanakos, MD, PhD, Principal Investigator — Department of Neurosurgery, Olympion Medical Center, 26443, Patras, GREECE
Locations (1):
- Olympion Medical Center, Pátrai, Greece

REFERENCES:
- [Derived] Karamanakos PN. Possible role for furazolidone in the treatment of glioblastoma multiforme. J BUON. 2013 Oct-Dec;18(4):1097. No abstract available. PMID 24344045